CLINICAL TRIAL: NCT05305417
Title: Cell-free Autologous Regenerative Endodontics Treatment for Permanent Mature Teeth With Pulp Necrosis and Periapical Lesions: a Randomized, Controlled Phase III Clinical Trial (CARETT)
Brief Title: Cell-free Autologous Regenerative Endodontics Treatment for Teeth With Periapical Lesions (CARETT)
Acronym: CARETT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 211
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Periapical Diseases; Pulp Necroses
Keywords: Regenerative Endodontics; Permanent Dentition; Pulp Necroses; Periapical Diseases; Root Canal Filling Material
MeSH Terms: conditions — Periapical Diseases; Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants don´t know wich intervention receive Investigator (outcome evaluator) don´t know wich intervention evaluate Outcomes Assessor (statistics) don´t know wich arm data evaluate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regenerative Endodontic Treatment (Experimental): This treatment consists of obturated the root canal preparations under an biological-based protocol using autologous biological elements and bioactive materials that allows restore the connective pulp-like tissue within the canals.
  Interventions: Procedure: Autologous Regenerative Endodontic Treatment
- Conventional root canal treatment (Active Comparator): This treatment consist on obturated the root canal preparations under the conventional protocol with an inert biomaterials like guttapercha and endodontics cements to seal the root canals.
  Interventions: Procedure: Conventional Root Canal Treatment

INTERVENTIONS:
Procedure: Autologous Regenerative Endodontic Treatment — The intervention consist in achieve an access to the teeth root canal system, do a chemico-mechanical preparation each root canal for to be obturated with an autologous biological scaffold and bioactive biomaterials to maintain teeth free of signs/symptoms caused by pulp necroses and periapical lesions
  Other Names: Pulp revascularization; Pulp revitalization; Pulp regeneration
  Arms: Regenerative Endodontic Treatment
Procedure: Conventional Root Canal Treatment — The intervention consist in achieve an access to the teeth root canal system, do a chemico-mechanical preparation each root canal for to be obturated with an inert biomaterial to maintain teeth free of signs/symptoms caused by pulp necroses and periapical lesions
  Other Names: Endodontically-treated Teeth
  Arms: Conventional root canal treatment

SUMMARY:
Conventional endodontic treatment has been the treatment of choice for the management of signs and symptoms of mature permanent teeth with pulpal necrosis and periapical lesion with predictable and favorable results. However, treatment outcomes have not shown improvement or innovation in decades. The main objective of this study is to evaluate the clinical effectiveness of a regenerative endodontic procedure (cell-free and autologous protocol) versus conventional endodontics in the resolution of signs and symptoms of periapical lesion and pulp vitality-sensitivity in mature permanent teeth with a diagnosis of pulpal necrosis and periapical lesion.

DETAILED DESCRIPTION:
Conventional endodontic treatment has been an effective treatment option for decades to treat signs and symptoms in mature permanent teeth with a diagnosis of apical lesion due to pulpal necrosis, allowing the teeth to be kept in the mouth free of signs/symptoms but devitalized. The clinical effectiveness of conventional treatment in this type of case is ≥80%, with some variations according to different studies. Despite advances and modifications in treatment protocols, this therapy has not shown improvements or innovations in its results in recent decades. The Regenerative Endodontics alternative is postulated as a biologically based endodontic treatment option that allows to resolve the signs and symptoms along with dental revitalization through the regeneration of the pulpal connective tissue, generating a substantive possibility of innovation and improvements to the therapy of conventional endodontics.

Various regenerative endodontic protocols have been proposed to achieve pulp tissue regeneration, from sophisticated techniques that involve cell transplantation, provision of scaffolds and/or signaling molecules, or simpler protocols that appeal to the autologous capacity of the organism to regenerate tissue. lost.

The main objective of this study is to evaluate the clinical effectiveness of a cell-free regenerative endodontic procedure with the contribution of an autologous scaffold (L-PRF) versus conventional endodontics in the recovery of signs of periapical lesion and pulp vitality-sensitivity in mature permanent teeth with diagnosis of pulpal necrosis and periapical lesion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (18-60y) systemically healthy or chronic disease controlled
* Uniradicular or multiradicular permanent mature teeth
* Teeth with diagnosis of pulp necrosis (negative response to thermal-cold pulp test) and sings or symptoms (clinical-radiographic) of periapical lesion.
* Root anatomy with curvatures ≤ 30°
* Feasibility of adhesive tooth restoration (direct or indirect)
* Voluntary participation under informed consent

Exclusion Criteria:

* Pregnant or lactating woman
* Signs of moderate or severe periodontal disease
* Teeth with signs of radicular fracture (vertical or horizontal), signs of root resorption (endo-exo)
* teeth with impossibility of good prognosis of coronary rehabilitation by direct or indirect adhesive technique
* Teeth that to treat can not to be correctly isolate with rubber dam

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of therapy | 12 month
  Number of treated tooth that remain in mouth free of clinical (negative percussion, negative palpation, abscence of inflammation, pain and fistula) and radiographic (total or partial reduction on size of periapical lesion) signs or symptoms at 12 month post operatory.

SECONDARY OUTCOMES:
Tooth re-sensibilization | 3, 6 and 12 month
  Number of treated tooth that response positively to thermal pulp sensibility test (cold stimulus) after 3, 6 and 12 months post operatory in relation with the initial negative pulp test. The positive-negative pulp sensibility response of treated teeth first is standardized testing the homologous vital tooth on the mouth.
Tooth re-vitalization | 3, 6 and 12 month
  Number of treated tooth that response positively to Vitality Pulp Test Doppler laser flowmetry after 3, 6 and 12 month. This Vitality Test assess pulpal blood flow by the detection of light scatter generated by moving erythrocytes. The positive-negative pulp vitality response of the treated teeth first is standardized testing the homologous vital tooth on the mouth.
Periapical lesion resolution | 3, 6 and 12 month
  Resolution of an periapical lesion using Periapical Index (PI), a scoring system for registration of apical periodontitis in radiographs
Procedure Time | intraoperatory
  total time required to perform each of the therapies recorded in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Caro, MSC, DDS, Study Director — Department of Endodontics, Faculty of Dentistry, University of Valparaíso, Chile.; Juan Caro, DDS, Principal Investigator — Department of Endodontics, Faculty of Dentistry, University of Valparaíso, Chile.

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: from start of participants recruitment to 12 months after publication of results
Access Criteria: The IPD data will be shared with any colleague or researcher that solicited the information by email to principal investigator explaining clear and direct the academic or research intention use of the data

REFERENCES:
- [Background] Glynis A, Foschi F, Kefalou I, Koletsi D, Tzanetakis GN. Regenerative Endodontic Procedures for the Treatment of Necrotic Mature Teeth with Apical Periodontitis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. J Endod. 2021 Jun;47(6):873-882. doi: 10.1016/j.joen.2021.03.015. Epub 2021 Mar 31. PMID 33811981
- [Background] Marquis VL, Dao T, Farzaneh M, Abitbol S, Friedman S. Treatment outcome in endodontics: the Toronto Study. Phase III: initial treatment. J Endod. 2006 Apr;32(4):299-306. doi: 10.1016/j.joen.2005.10.050. PMID 16554199
- [Background] Friedman S, Abitbol S, Lawrence HP. Treatment outcome in endodontics: the Toronto Study. Phase 1: initial treatment. J Endod. 2003 Dec;29(12):787-93. doi: 10.1097/00004770-200312000-00001. PMID 14686806
- [Background] Farzaneh M, Abitbol S, Lawrence HP, Friedman S; Toronto Study. Treatment outcome in endodontics-the Toronto Study. Phase II: initial treatment. J Endod. 2004 May;30(5):302-9. doi: 10.1097/00004770-200405000-00002. PMID 15107640
- [Background] Moazami F, Sahebi S, Sobhnamayan F, Alipour A. Success rate of nonsurgical endodontic treatment of nonvital teeth with variable periradicular lesions. Iran Endod J. 2011 Summer;6(3):119-24. Epub 2011 Aug 15. PMID 23130063
- [Background] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729
- [Background] Ng YL, Mann V, Rahbaran S, Lewsey J, Gulabivala K. Outcome of primary root canal treatment: systematic review of the literature -- Part 2. Influence of clinical factors. Int Endod J. 2008 Jan;41(1):6-31. doi: 10.1111/j.1365-2591.2007.01323.x. Epub 2007 Oct 10. PMID 17931388
- [Background] Ng YL, Mann V, Rahbaran S, Lewsey J, Gulabivala K. Outcome of primary root canal treatment: systematic review of the literature - part 1. Effects of study characteristics on probability of success. Int Endod J. 2007 Dec;40(12):921-39. doi: 10.1111/j.1365-2591.2007.01322.x. Epub 2007 Oct 10. PMID 17931389
- [Background] Diogenes A, Ruparel NB. Regenerative Endodontic Procedures: Clinical Outcomes. Dent Clin North Am. 2017 Jan;61(1):111-125. doi: 10.1016/j.cden.2016.08.004. PMID 27912813
- [Background] Widbiller M, Eidt A, Lindner SR, Hiller KA, Schweikl H, Buchalla W, Galler KM. Dentine matrix proteins: isolation and effects on human pulp cells. Int Endod J. 2018 May;51 Suppl 4:e278-e290. doi: 10.1111/iej.12754. Epub 2017 Mar 14. PMID 28211068
- [Background] Galler KM, Buchalla W, Hiller KA, Federlin M, Eidt A, Schiefersteiner M, Schmalz G. Influence of root canal disinfectants on growth factor release from dentin. J Endod. 2015 Mar;41(3):363-8. doi: 10.1016/j.joen.2014.11.021. Epub 2015 Jan 13. PMID 25595468
- [Background] Galler KM, D'Souza RN, Federlin M, Cavender AC, Hartgerink JD, Hecker S, Schmalz G. Dentin conditioning codetermines cell fate in regenerative endodontics. J Endod. 2011 Nov;37(11):1536-41. doi: 10.1016/j.joen.2011.08.027. PMID 22000458
- [Background] Smith AJ, Scheven BA, Takahashi Y, Ferracane JL, Shelton RM, Cooper PR. Dentine as a bioactive extracellular matrix. Arch Oral Biol. 2012 Feb;57(2):109-21. doi: 10.1016/j.archoralbio.2011.07.008. PMID 21855856
- [Background] Galler KM. Clinical procedures for revitalization: current knowledge and considerations. Int Endod J. 2016 Oct;49(10):926-36. doi: 10.1111/iej.12606. Epub 2016 Feb 1. PMID 26715631
- [Background] Ducret M, Fabre H, Celle A, Mallein-Gerin F, Perrier-Groult E, Alliot-Licht B, Farges JC. Current challenges in human tooth revitalization. Biomed Mater Eng. 2017;28(s1):S159-S168. doi: 10.3233/BME-171637. PMID 28372291
- [Background] Chrepa V, Henry MA, Daniel BJ, Diogenes A. Delivery of Apical Mesenchymal Stem Cells into Root Canals of Mature Teeth. J Dent Res. 2015 Dec;94(12):1653-9. doi: 10.1177/0022034515596527. Epub 2015 Jul 20. PMID 26195498
- [Background] Arslan H, Ahmed HMA, Sahin Y, Doganay Yildiz E, Gundogdu EC, Guven Y, Khalilov R. Regenerative Endodontic Procedures in Necrotic Mature Teeth with Periapical Radiolucencies: A Preliminary Randomized Clinical Study. J Endod. 2019 Jul;45(7):863-872. doi: 10.1016/j.joen.2019.04.005. Epub 2019 May 31. PMID 31155298
- [Background] Jha P, Virdi MS, Nain S. A Regenerative Approach for Root Canal Treatment of Mature Permanent Teeth: Comparative Evaluation with 18 Months Follow-up. Int J Clin Pediatr Dent. 2019 May-Jun;12(3):182-188. doi: 10.5005/jp-journals-10005-1616. PMID 31708612
- [Background] Brizuela C, Meza G, Urrejola D, Quezada MA, Concha G, Ramirez V, Angelopoulos I, Cadiz MI, Tapia-Limonchi R, Khoury M. Cell-Based Regenerative Endodontics for Treatment of Periapical Lesions: A Randomized, Controlled Phase I/II Clinical Trial. J Dent Res. 2020 May;99(5):523-529. doi: 10.1177/0022034520913242. Epub 2020 Mar 23. PMID 32202965
- [Background] About I. Proceedings of the Pulp Biology and Regeneration Group Symposium 2019: Bridging Basic and Translational Research in Pulp Biology-Developing Technologies for Regenerating Vital Dental Tissues. J Endod. 2020 Sep;46(9S):S1. doi: 10.1016/j.joen.2020.06.018. No abstract available. PMID 32950179
- [Background] He L, Kim SG, Gong Q, Zhong J, Wang S, Zhou X, Ye L, Ling J, Mao JJ. Regenerative Endodontics for Adult Patients. J Endod. 2017 Sep;43(9S):S57-S64. doi: 10.1016/j.joen.2017.06.012. PMID 28844305